CLINICAL TRIAL: NCT02502565
Title: Musculoskeletal Ultrasound in Asymptomatic Hyperuricemia: Redefining Early Urate Disease
Brief Title: Musculoskeletal Ultrasound in Asymptomatic Hyperuricemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Howard University (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: MIRB #01580
Record Dates: First submitted 2015-06-24; First posted 2015-07-20 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Uric Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Uric Acid Level
  Interventions: Other: Uric acid level

INTERVENTIONS:
Other: Uric acid level

SUMMARY:
An observational study to evaluate the prevalence of US changes of gout in the joints and tendons of patients with different degrees of asymptomatic hyperuricemia. The investigators' findings may support the extension of the spectrum of urate disease, and define a subset of patients that may benefit from early urate-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have at least one serum uric acid level l ≥ 7.0 mg/dL within the last two years without a clinical diagnosis of gout per American College of Rheumatology criteria30 (appendix A).
2. Patients, of matched gender and age, with normal uric acid levels will serve as controls.

Exclusion Criteria:

1. Patients who meet or have met the ACR criteria for Gout, unable to read English, and/or have terminal illness will not be eligible to participate in the study.
2. Patients with a diagnosis of skin psoriasis31, rheumatoid arthritis, or spondyloarthropathies will not be eligible to participate.
3. Patients who are on urate-lowering therapy.
4. Patients with 1 or 2 total knee replacements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: US Veterans with asymptomatic hyperuricemia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of Urate Depositions Detected in Ultrasound | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gail S Kerr, MD, FRCP, Principal Investigator — Washington VAMC
Locations (2):
- United States (2):
  - Howard University Hospital, Washington D.C., District of Columbia
  - WashingtonVAMC, Washington D.C., District of Columbia